CLINICAL TRIAL: NCT00089466
Title: Phase IB/IIA Dose-Finding Safety and Activity Study of AMD11070 (An Orally Administered CXCR4 Entry Inhibitor) in HIV-Infected Subjects
Brief Title: Safety and Activity of the Oral HIV Entry Inhibitor AMD11070 in HIV Infected Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Advancing Clinical Therapeutics Globally for HIV/AIDS and Other Infections (Network)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A5210; 10020 (Registry Identifier: DAIDS ES); ACTG A5210
Record Dates: First submitted 2004-08-05; First posted 2004-08-06 (Estimated); Last update posted 2021-11-09 (Actual); Status verified 2012-10

CONDITIONS: HIV Infections
Keywords: Entry Inhibitors; CXCR4 Entry Inhibitors; Treatment Experienced; Treatment Naive
MeSH Terms: conditions — HIV Infections | interventions — mavorixafor

ARMS (8):
- A (Experimental): 200 mg AMD11070 every 12 hours
  Interventions: Drug: AMD11070
- B (Experimental): 400 mg AMD11070 every 12 hours
  Interventions: Drug: AMD11070
- C (Experimental): 600 mg AMD11070 every 12 hours
  Interventions: Drug: AMD11070
- D (Experimental): 800 mg AMD11070 every 12 hours
  Interventions: Drug: AMD11070
- E (Experimental): 1000 mg AMD11070 daily
  Interventions: Drug: AMD11070
- F (Experimental): 1500 mg AMD11070 daily
  Interventions: Drug: AMD11070
- G (Experimental): 1000 mg AMD11070 every 12 hours
  Interventions: Drug: AMD11070
- H (Experimental): 2000 mg AMD11070 daily
  Interventions: Drug: AMD11070

INTERVENTIONS:
Drug: AMD11070 — AMD11070 taken daily. Dosage dependent on arm.

SUMMARY:
New treatment options are critical for treatment-experienced HIV infected patients with drug resistance. HIV entry inhibitors have been shown effective in patients with resistance to other anti-HIV drugs. This study will test the safety and anti-HIV activity of eight different doses of the HIV entry inhibitor AMD11070 (also known as AMD070) in HIV infected patients.

DETAILED DESCRIPTION:
AMD11070 is an oral HIV-1 entry inhibitor that targets the CXCR4 receptor on T cells. AMD11070 has been shown safe and well-tolerated in Phase I clinical trials in HIV uninfected people. The goal of this study is to evaluate the safety and antiretroviral activity of eight dose levels of AMD11070 in HIV infected adults with X4-tropic virus. Pharmacokinetics (PK) of AMD11070 will also be studied.

This study will last 90 days. All participants will receive medication for 10 days. There are eight cohorts in this study, with a maximum of six participants per cohort. Cohort A will receive 200 mg AMD11070 every 12 hours; Cohort B will receive 400 mg AMD11070 every 12 hours; Cohort C will receive 600 mg AMD11070 every 12 hours; Cohort D will receive 800 mg AMD11070 every 12 hours; Cohort E will receive 1000 mg AMD11070 daily; Cohort F will receive 1500 mg AMD11070 daily; Cohort G will receive 1000 mg AMD11070 every 12 hours; and Cohort H will receive 2000 mg AMD11070 daily. Cohorts B, C, D, and E will open sequentially, provided no more than one of six participants in the preceding cohort experiences dose-limiting toxicity (DLT) based on safety evaluations through Day 17. Cohort G will open to enrollment when Cohort E is filled; Cohort H will open to enrollment when Cohort F is filled. Cohort F will open to enrollment provided no more than one of six participants of Cohorts E and G experiences DLT. All study participants will be offered to receive open-label AMD11070 through a separate long-term safety study.

Participants will either be admitted to the general clinical research center (GCRC) for the dosing period or have dosing, PK testing, and other study monitoring done on an outpatient basis, depending on the study site. Participants admitted to the GCRC for the dosing period will be allowed daytime passes from the GCRC on Days 4, 6, 7, 8, and 9. During the study, participants will have continuous heart monitoring, serial electrocardiograms (EKGs), and vital sign checks. Fasting blood collection will occur on Days 5 and 10. Trough PK testing will occur at entry and on Days 1, 2, 3, 4, 6, 8, and 11. Intensive 24-hour PK testing and 24-hour urine collection will occur on Days 10 and 11. After treatment, targeted physicals and urine collection will occur on Days 17, 30, and 90, and additional blood collection will occur on Days 17, 21, 30, and 90. Participants will undergo an EKG on Days 17 and 90. Participants will also undergo an opthalmologic evaluation and questionnaire sometime after receiving AMD11070.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infected
* Have X4- or dual/mixed-tropic virus confirmed no more than 56 days prior to study entry
* HIV-1 viral load of 5,000 copies/ml or more within 60 days prior to study entry
* If female, willing to discontinue hormonal contraception 1 week prior to study entry
* Willing to use acceptable forms of contraception

Exclusion Criteria:

* Antiretroviral treatment within 14 days prior to study entry
* Other prescription medications, herbal supplements, or aspirin within 7 days prior to study entry. Patients taking medication for prophylaxis for Pneumocystis carinii pneumonia (PCP) are not excluded. Patients taking medications approved by protocol officials are not excluded, provided they have been on a stable dose for at least 14 days prior to study entry.
* Nonsteroidal anti-inflammatory drugs (NSAIDS), over the counter medications, or other supplements (including multivitamins) within 1 day prior to study entry
* Heavy exercise within 24 hours before study entry evaluations are done
* Immunizations within 30 days prior to study entry
* Radiation therapy, cytotoxic chemotherapeutic agents, or immunomodulatory agents within 30 days prior to study entry
* Current use of some CYP substrates, inhibitors, or inducers. Use of CYP450 substrates is allowed, except for CYP2D6 and CYP2C8 substrates.
* Current use of P-gp inducers or inhibitors
* Allergy or sensitivity to study drug or its formulations
* Active infection or acute illness within 14 days prior to study entry, including HIV-associated opportunistic infections
* History of heart abnormalities. Patients with any repolarization delay (QTc interval of greater than 500 msec) or a history of additional risk factors for torsade de pointes (e.g., heart failure, hypokalemia) are also excluded.
* Drug or alcohol abuse or dependence or other medical or psychological condition that, in the opinion of the investigator, would interfere with the study or put participants at undue risk
* Chronic diarrhea, defined as having more than 3 stools/day for more than 4 weeks prior to study entry
* Pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2004-11; Primary Completion 2006-06 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicities of Grade 3 or greater | during the 10 days of treatment or the 7 days after stopping treatment
Reduction in X4-tropic virus from baseline of 1 log10 relative luciferase units (rlu) | day 10

CONTACTS AND LOCATIONS:
Overall Officials: Michael S. Saag, MD, Study Chair — University of Alabama at Birmingham
Locations (3):
- United States (3):
  - Alabama Therapeutics CRS, Birmingham, Alabama
  - The Ponce de Leon Ctr. CRS, Atlanta, Georgia
  - Indiana Univ. School of Medicine, Infectious Disease Research Clinic, Indianapolis, Indiana

REFERENCES:
- [Background] De Clercq E. Emerging anti-HIV drugs. Expert Opin Emerg Drugs. 2005 May;10(2):241-73. doi: 10.1517/14728214.10.2.241. PMID 15934866
- [Background] Moore JP, Kitchen SG, Pugach P, Zack JA. The CCR5 and CXCR4 coreceptors--central to understanding the transmission and pathogenesis of human immunodeficiency virus type 1 infection. AIDS Res Hum Retroviruses. 2004 Jan;20(1):111-26. doi: 10.1089/088922204322749567. PMID 15000703
- [Background] Reeves JD, Piefer AJ. Emerging drug targets for antiretroviral therapy. Drugs. 2005;65(13):1747-66. doi: 10.2165/00003495-200565130-00002. PMID 16114975
- [Background] Ruibal-Ares BH, Belmonte L, Bare PC, Parodi CM, Massud I, de Bracco MM. HIV-1 infection and chemokine receptor modulation. Curr HIV Res. 2004 Jan;2(1):39-50. doi: 10.2174/1570162043484997. PMID 15053339
- [Background] Shaheen F, Collman RG. Co-receptor antagonists as HIV-1 entry inhibitors. Curr Opin Infect Dis. 2004 Feb;17(1):7-16. doi: 10.1097/00001432-200402000-00003. PMID 15090884